CLINICAL TRIAL: NCT00920894
Title: The Effect of Plant Stanol Esters on Serum Total and Lipoproteins Lipids, Non-cholesterol Sterols and Apolipoproteins in Subjects With Elevated Blood Lipid Concentration
Brief Title: Effect of Plant Stanol Esters on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Life Sciences Ltd. (Other)
Responsible Party: Päivi Cheney, MD, Clinical Life Sciences Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kainuu PlantStanol Ester Study
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Elevated Blood Lipids
MeSH Terms: interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- yoghurt type minidrink containing plant stanol ester (Experimental)
  Interventions: Dietary Supplement: plant stanol ester
- yoghurt type minidrink without plant stanol ester (Placebo Comparator)
  Interventions: Dietary Supplement: plant stanol ester

INTERVENTIONS:
Dietary Supplement: plant stanol ester — the effect of plant stanol esters on plasma lipids

SUMMARY:
This study aims to measure the effect of plant stanol esters on serum total and lipoproteins lipids, non-cholesterol sterols and apolipoproteins in subjects with elevated fasting blood lipid concentrations

DETAILED DESCRIPTION:
The link between high serum low-density lipoprotein (LDL) cholesterol and cardiovascular disease has long been recognized. Dietary plant stanol esters have been shown to effectively reduce serum levels of total and LDL cholesterol. Plant stanols decrease the absorption of both biliary and dietary cholesterol from the small intestine and thereby reduce serum LDL cholesterol levels.

This study aims to verify the effect of plant stanol esters on blood lipids. Subjects with elevated fasting blood lipid concentrations will be randomized to study groups. The groups consume yoghurt type minidrink containing plant stanol ester (2 g plant stanols per day) or similar minidrink without plant stanol esters. After 10 weeks study period serum total and lipoproteins lipids, non-cholesterol sterols and apolipoproteins will by analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood lipids
* Body Mass Index < 35 kg/m2
* Stable body weight

Exclusion Criteria:

* Receiving medications or supplements other than stable statin therapy known to affect lipid metabolism
* Severe obesity
* Hyperglycemia
* Severe diseases (inc. diabetes, unstable CVD, malignant disease, inflammatory disease, gastrointestinal disease)
* Hepatic, kidney or thyroid disease or disorder
* Pregnancy or breast feeding
* Severe intolerance or allergy to any ingredient of test product

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
plasma lipids | 10 weeks

SECONDARY OUTCOMES:
plasma lipoprotein lipids non-cholesterol sterols | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Life Sciences Ltd, Vuokatti, Finland